CLINICAL TRIAL: NCT05176444
Title: Managing the Needs of Care Home Residents Through a Music Therapy Intervention: A Non-randomised Feasibility Trial
Brief Title: Managing the Needs of Care Home Residents With Dementia Through a Music Therapy Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anglia Ruskin University (Other)
Collaborators: Anchor Trust (Other); The Utley Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U4-11662
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cognitive Impairment; Dementia
Keywords: Dementia; Music therapy; Cognition; Care home; Quality of care; Non-pharmacological intervention; Needs; Neuropsychiatric symptoms
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy intervention (Experimental): Music therapy
  Interventions: Behavioral: Music therapy
- Control group - standard care (No Intervention): Standard care for residents with cognitive impairment. Staff will not receive music therapy training.

INTERVENTIONS:
Behavioral: Music therapy — Individual music therapy sessions across 12-weeks with people with cognitive impairment/dementia. Music therapy training for care home staff at four time points across 12-weeks.
  Arms: Music therapy intervention

SUMMARY:
The purpose of this study is to implement and evaluate a music therapy intervention in care homes. The primary aim is to assess whether implementing the intervention will have an impact on unmet in care homes for people living with dementia. Researchers will also examine the feasibility of a music therapy programme in care homes and its effects on care staff and residents with cognitive impairment. Care home staff will also receive training with music therapists via video communications to help staff use music therapy techniques to support people living with dementia.

DETAILED DESCRIPTION:
This project aims to evaluate the feasibility and effectiveness of a 12-week music therapy programme in care homes for residents with cognitive impairment/dementia and care home staff using a non-randomised control design. Music therapy is widely recognised as beneficial for people living with dementia. However, little is known about its overall impact on quality of care in care homes.

Research questions:

1. Can a music therapy intervention improve quality of care in care homes by supporting residents' needs?
2. What are the effects of music therapy on residents with cognitive impairment and care home staff?
3. Is the implementation of a music therapy programme feasible in care homes?
4. For the treatment of symptoms of dementia, is music therapy a cost-effective treatment in care homes?

Intervention:

The team will invite a total of 84 participants from 12 care homes located across the North and South of England to take part in the study. This includes 48 participants with cognitive impairment/dementia and 36 care home staff. The team will recruit a qualified music therapist in each region to work within the care home to deliver the music therapy intervention.

Residents with cognitive impairment/dementia will be invited to receive twenty 30-minute individual music therapy sessions across 12 weeks. The therapy will be video recorded for training purposes. Data will be collected about residents to learn about their needs and any health and wellbeing symptoms. This will help inform music therapists about each individuals' specific needs so that they can tailor a suitable treatment approach. They will enable a meaningful, engaging therapeutic relationship to improve the health and wellbeing of residents. The sessions will focus on targeting specific behavioural and psychological symptoms of dementia by providing cognitive stimulation, communicative support and social connectedness.

Within the 12-week programme, care home staff participants will be invited to collectively receive music therapy training on four occasions during week 3, 6, 9 and 12. Each music therapist will demonstrate significant moments of their sessions to staff via short video clips from a music therapy session. They will provide clinical explanations to staff about the techniques they have used and why they are effective for the individuals with cognitive impairment.

Data collection:

The team will be collecting a range of qualitative and quantitative data. The researchers will use an integrated evaluative approach focussing on clinical and organisational outcomes to examine the research questions. As part of the non-randomised control design, six of the care homes will be in the intervention group and receive the music therapy programme. There will be 42 participants in this group (24 with cognitive impairment, 18 care home staff). The remaining six care homes will form the control group and receive treatment as usual. Baseline and post 12-week data will be collected from all homes to compare differences between groups. Within group data will also be compared from the intervention homes.

Once all of the data has been collected from the control group care homes, they will then go on to receive the music therapy programme with the same amount and ratio of participants.

Implications:

The study has the potential to improve the lives of care home residents living with cognitive impairment/dementia. It also has the potential to improve the work life of care home staff and generate better quality of care. Staff will be provided with the tools and understanding of music therapy techniques, so that the potential effects can be sustainable. Standardised protocols are needed to learn about how researchers and practitioners can work with the social care sector to implement an effective music therapy programme. The evaluation of this study will inform this sector about the feasibility and effectiveness of music therapy care in care homes. The study findings will provide valuable insights into how to transform the social care sector through psychosocial, non-pharmacological intervention at micro and macro level.

.

ELIGIBILITY:
Inclusion criteria

The proposed inclusion criteria for care home residents are as follows:

* Participants must be aged 50+ years
* Participants will be a resident of one of the 12 care homes taking part
* For each participant, there must be clinical evidence of cognitive impairment. This will be determined by a score of 24 or under on the SMMSE
* Each participant must display at least one behavioural/psychological symptom of dementia. This will be determined by a score of 4 or higher on the NPI-NH.

The proposed inclusion criteria for care home staff are as follows:

* Participants must be aged 18+ years
* Participants must have worked in the care home for at least 3 months
* Participants will be required to have in-depth knowledge of the resident participant(s). This will be determined through communications with home managers to ensure each staff member is paired with a resident they provide regular care for.

Exclusion Criteria

Exclusion criteria for care home residents:

- Participants who's health appears to be at risk which raises the concerns of their sustained involvement with the study. This would be evident from a health assessment from a general practitioner. Given that this is a music therapy study, this could also include people with a hearing impairment.

Exclusion criteria for care home staff:

- Staff who cannot adequately answer on behalf of the residents due to lack of knowledge of the residents.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Camberwell Assessment of Needs in the Elderly - CANE | 15 minutes
  For people with cognitive impairment - to measure the quality of care in care homes by assessing individual needs. This measure examines met and unmet needs in older people in 24 areas from self-care to communicative abilities. 1 = a met need, 2 = an unmet need. Met needs and unmet needs are totalled. A higher score indicates a higher number of needs.

SECONDARY OUTCOMES:
Standardised Mini Mental State Examination - SMMSE | 15 minutes
  For people with cognitive impairment - a standardised assessment to test cognitive function of residents in care homes. This version will factor in participants with various impairments such as visual and motor issues. Scores are between 0 and 30. Lower scores indicate lower cognitive function.
Neuropsychiatric Inventory Nursing Homes - NPI-NH | 12 minutes
  Care home staff will be interviewed to measure the neuropsychiatric symptoms of people with dementia in care homes. Data is collected about a range of symptoms from A-J including delusions, anxiety, aberrant motor behaviours, disinhibition. If a symptom is present, the frequency is scored from 1 (rarely) - 4 (very often), the severity is scored from 1 (mild) - 3 (severe). Frequency x severity provides an NPI score for each present symptom which is totalled. Occupational disruptiveness is also scored for a present symptom from 1 (not at all) - 5 (very severe). Occupational disruptiveness scores are totalled to provide an overall score.
EuroQoL - EQ-5D-5L - self completion | 5 minutes
  Residents will respond to which level they perceive in five domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with level 1 (no problem) to level 5 (extremely). Each number representing a level will develop a code (e.g. 11111 would indicate no problems in health related quality of life). These scores can then be formulated into an index value.
EuroQoL - EQ-5D-5L - proxy | 5 minutes
  The same measure as above to assess proxy health related quality of life. This will be completed by a care staff member and scoring will be as above.
Barthel Index (BI) | 10 minutes
  A survey link will be sent out to care staff to measure the perceived functional abilities of the individuals with dementia such as feeding, bathing etc. Care staff will be asked the questions to provide their opinions on one domain (activities of daily living) with 10 items. Scores range between 0 and 100. A higher score indicates a better outcome with higher levels of independence.
Job Satisfaction Index (JSI) | 10 minutes
  A survey link will be sent out to care staff to measure job satisfaction based on 18 statements using five categories from strongly agree - strongly disagree.
Maslach Burnout Inventory - Human services (MBI-HSS) | 10 minutes
  A survey link will be sent out to care staff to measure burnout. Questions are based around three areas: emotional exhaustion, depersonalisation and personal accomplishments. There are a total of 22 questions related to how one feels in their job, on a scale from 0 (never) - 6 (every day). Average scores are calculated.
Qualitative semi-structured Interviews | 10 - 20 minutes
  A semi-structured interview with care staff will be carried out at baseline in both groups until data saturation is met. This interview consists of questions about the concept of quality of care and job satisfaction. Another interview will be carried out with all care staff participants in the intervention group at the end of the music therapy treatment to evaluate the music therapy process.
Client Service Receipt Inventory (CSRI Dementia) | 15 minutes
  A measure of the cost effectiveness of the music therapy in care homes. This instrument collects information about service usage of residents, medication usage and overall care home costs.
Total number of staff at the care home | 2 minutes
  The total number of staff at each care home is collected in both groups, pre and post to examine staff retention and turnover.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Odell-Miller, PhD, Study Director — Anglia Ruskin University
Locations (11):
- United Kingdom (11):
  - Ridgemount, Banstead, Surrey
  - Oakleigh, Godstone, London, Surrey
  - Greenacres, Banstead, London, Surrey
  - Hatfield House, Doncaster
  - Simon Marks Court, Leeds
  - Oak Tree Lodge, Leeds
  - Kimberly Court, Newquay
  - Wharfside, Otley
  - St Anne's, Saltash
  - Prior Bank, Sheffield
  - Herries Lodge, Sheffield

IPD SHARING:
Plan to Share IPD: No
Data will be anonymous

REFERENCES:
- See also: This study has tested similar methods to those that are being used in the current study — https://bmcgeriatr.biomedcentral.com/articles/10.1186/s12877-015-0082-4
- See also: This study has informed the current study of outcome measures to use — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5491018/
- See also: This study details the effects of music therapy on dementia and highlights the need for further trials — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7248378/